CLINICAL TRIAL: NCT04974125
Title: Drain-Exsu: Phase III Trial Assessing the Effect of Peritoneal Gas Drain on Postoperative Pain in Gynecologic Minimally Invasive Surgery
Brief Title: Impact of Peritoneal Gas Drain on Postoperative Pain for Gynaecological Cancer Patients With Minimally Invasive Surgery
Acronym: DRAIN-EXSU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Oscar Lambret (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: DRAIN-EXSU-1907
Record Dates: First submitted 2021-05-06; First posted 2021-07-23 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Gynaecologic Cancer
Keywords: Postoperative pain; Peritoneal gas drainage; Laparoscopic gynaecological surgery; Robotised laparoscopic gynaecological surgery
MeSH Terms: conditions — Pain, Postoperative | interventions — Drainage

STUDY DESIGN:
Intervention Model Description: Patient will be pre-selected before medical operation. During the surgery, if the surgeon performs only the laparoscopy, the patient will be randomized. Then, the allocated procedure (with or without drain) will be carried out.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A :Aspiration of peritoneal gas through a drain (Experimental): Patients in experimental arm will receive surgery (either laparoscopic or robotised laparoscopic surgery). The exsufflation will be carrying out by a drain.
  Then, patients will be followed-up during 7 days after surgery.
  Interventions: Procedure: Drain
- Arm B : Manual evacuation of the peritoneal gas, via the trocar (Active Comparator): Laparoscopic or robotised laparoscopic surgery + Trocar
  Patient in this experimental arm will receive surgery (either laparoscopic or robotised laparoscopic surgery). The exsufflation will be carrying out carried out manually using the trocar (standard of care).Then, patient will be followed-up during 7 days after surgery.
  Interventions: Procedure: Manual exsufflation

INTERVENTIONS:
Procedure: Drain — A 10 mm suction drain is placed through a trocar in the right hypochondrium (liver).
  Arms: Arm A :Aspiration of peritoneal gas through a drain
Procedure: Manual exsufflation — Exsufflation through the trocar opening.
  Arms: Arm B : Manual evacuation of the peritoneal gas, via the trocar

SUMMARY:
This is a phase III, monocenter and randomized study, which evaluates the effectiveness of peritoneal gas drainage on postoperative pain in laparoscopic or robotic laparoscopic gynaecological surgery. This study aim is to assess the efficacy of active gas extraction with a drain (arm A) in comparison to manual evacuation (arm B,) in terms of pain incidence reduction linked to laparoscopic or robotic laparoscopic surgery.

DETAILED DESCRIPTION:
The primary objective is to assess the efficacy of active gas aspiration compared to simple manual gas evacuation to reduce the incidence of specific laparoscopic surgery pain.

Secondary objectives of this study include :

* Comparing the evolution of specific pains after laparoscopic surgery, between study groups
* Description of postoperative antalgics consumption in each group
* Evaluating the safety of the evaluated procedure
* Evaluating the impact of the evaluated procedure on hospitalisation duration ( for patients with ambulatory surgery initially planned)

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 ans ;
* Woman who underwent laparoscopic or robotised laparoscopic surgery in peritoneal cavity (benign or malignant gynaecological affection) ;
* Planned ambulatory surgery
* Patient willing and able to be treated and followed according the protocol during the trial ;
* Patient covered by the French "Social Security" regime ;
* Effective contraception for reproductive age patients ;
* Signed written informed consent before surgery

Per-operatory eligibility criterion :

* No conversion from laparoscopic surgery to laparotomy surgery

Exclusion Criteria:

* Extra-peritoneal surgery scheduled ( example : aortic dissection) ;
* Upper-abdomen surgery (example : liver, gall bladder) ;
* History of shoulders pains prior to surgery (the assessment must be carried out within a period of 30 days before the surgery) ;
* Inability to comply with medical follow-up of the trial (geographical, social or psychic reasons)
* Person under guardianship
* Pregnant or breastfeeding woman

Non eligibility criterion known during the operation :

* Conversion from laparoscopic surgery to laparotomy surgery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Gynaecological cancer
Enrollment: 202 (Actual)
Dates: Start 2022-01-07 (Actual); Primary Completion 2023-12-11 (Actual); Study Completion 2023-12-11 (Actual)

PRIMARY OUTCOMES:
Specific pain (shoulders and/or subcostal areas) related to the laparoscopic surgery (Day 0), measured with a numerical pain assessment scale (score from 0 to 10) | During the 24 hours after surgery
  Comparison on portion of patients with significative early pain linked to the laparoscopic surgery, between the two groups (Chi-2 tests).

SECONDARY OUTCOMES:
Maximal score pain, measured with a numerical pain assessment scale (score from 0 to 10) | 24 hours after surgery
  The maximum score pain will be evaluated by the mean difference between each group (Student or Mann-Whitney tests).
Assess pain at trocar holes comparatively in the two groups | 24 hours after surgery
  The site of pain will be reported to describe pain overall, but also specifically in the shoulders and/or subcostal areas and pain at trocar holes.
  Pain will be measured with the numerical pain assessment scale (score from 0 to 10).
Laparoscopic surgery specific pains, measured with a numerical pain assessment scale (score from 0 to 10) | 7 days after surgery
  A notebook filled in by the patient at home with a daily assessment of pain according to the numerical pain assessment scale, with a phone call from the nurse on day 7 (considering that the day of the surgery is day 0).
Antalgics consumption | 24 hours and 7 days after surgery
  Qualitative description through patient notebook.
Antalgics consumption | 24 hours and 7 days after surgery
  Quantitative description through patient notebook.
Adverse events (AE) (grade ≥III Clavien-Dindo classification) | 30 days after surgery
  Safety procedure will be describe through adverse events notification potentially related to the procedure and their grade (total amount of AE, maximal grade of AE per patient).
Evaluate the impact of the evaluated procedure on the hospitalisation duration | Through the study patient participation, an average of 2 months
  Impact of the peritoneal gas aspiration technique on the hospitalisation duration for patient with ambulatory surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Fabrice NARDUCCI, PhD, Study Director — Centre Oscar Lambret
Locations (1):
- Fabrice NARDUCCI, Lille, France